CLINICAL TRIAL: NCT04216823
Title: Evaluation of Perfusion Index as an Objective Measure for Supraclavicular Brachial Plexus Block in Pediatric Patients
Brief Title: Perfusion Index as an Objective Measure for Supraclavicular Brachial Plexus Block in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, aijun xu, associate professor, Tongji Hospital
Other Study IDs: PISP
Record Dates: First submitted 2019-12-28; First posted 2020-01-03 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Supraclavicular Brachial Plexus Block
Keywords: perfusion index; supraclavicular brachial plexus block; children
MeSH Terms: interventions — Perfusion Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sevoflurane Group: sevoflurane is used for anesthetic induction
  Interventions: Device: perfusion index
- Propofol Group: intravenous anesthetic propofol is used for anesthetic induction
  Interventions: Device: perfusion index

INTERVENTIONS:
Device: perfusion index — perfusion index in the prediction of peripheral block success was previously reported for infraclavicular brachial plexus block, axillary brachial plexus block, interscalene brachial plexus block, and supraclavicular brachial plexus in adult patients

SUMMARY:
The aim of the present study is to evaluate the effects of supraclavicular brachial plexus block using perfusion index in pediatric patients undergoing Upper limb surgery.

DETAILED DESCRIPTION:
The role of perfusion index in the prediction of peripheral block success was previously reported for infraclavicular brachial plexus block, axillary brachial plexus block, interscalene brachial plexus block, and supraclavicular brachial plexus in adult patients. The aim of the present study is to assess the effects of perfusion index on success of supraclavicular brachial plexus block in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* Children undergoing Upper limb surgery.
* Parents' agreement.

Exclusion Criteria:

* Parents' refusal.
* Children with behavioral changes
* Children with physical developmental delay
* Children on treatment with sedative or anticonvulsant.

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: ASA physical status I-II,Age 1 month-12 year,Children undergoing Upper limb surgery.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
perfusion index | the time span between 1 day preoperative and 24 hours after surgery
  Correlation between success of supraclavicular brachial plexus block and perfusion index

SECONDARY OUTCOMES:
mean arterial blood pressure | the time span between 1 day preoperative and 24 hours after surgery
  perioperative mean arterial blood pressure in mmHg
heart rate | the time span between 1 day preoperative and 24 hours after surgery
  perioperative heart rate as beat/min
PI ratio | up to 10 minutes
  Correlate between baseline PI and 10min after supraclavicular brachial plexus block

CONTACTS AND LOCATIONS:
Overall Officials: Hong Liu, Dr., Study Chair — Huazhong university, Tongji medical college
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chu T, Zhou S, Peng T, Tao H, Chen H, Yan X, Xin Y, Tian Z, Wang J, Deng L, Xu A. Perfusion Index Predicts the Effectiveness of Supraclavicular Brachial Plexus Block in Children Under General Anesthesia: A Randomized Controlled Trial. Anesthesiol Res Pract. 2025 Feb 22;2025:5583145. doi: 10.1155/anrp/5583145. eCollection 2025. PMID 40026611
- [Derived] Wang J, Deng L, Xu A. Evaluation of prediction effect of perfusion index for supraclavicular brachial plexus block in children: protocol for a randomized trial. Trials. 2022 Aug 4;23(1):629. doi: 10.1186/s13063-022-06597-y. PMID 35927745